CLINICAL TRIAL: NCT02514941
Title: Bioavailability of Paracetamol, Amoxicillin and Talinolol and Expression of Intestinal Drug Metabolizing Enzymes and Transport Proteins Before, Immediately and One Year After Proximal Roux-en-Y Gastric Bypass Operation in Patients With Morbid Adipositas
Brief Title: Bioavailability of Paracetamol, Amoxicillin and Talinolol Before, Immediately and One Year After Gastric Bypass Operation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Gastric Bypass
Record Dates: First submitted 2015-07-29; First posted 2015-08-04 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-07

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid | interventions — Acetaminophen; Amoxicillin; talinolol; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- pre OP (Experimental): The subjects will be administered 200 mg paracetamol, 250 mg amoxicillin and 50 mg talinolol dissolved in 40 ml water which must be drunken with additional 200 ml water on the first study day. This pharmacokinetic period will be performed within three days before the scheduled proximal Roux-en-Y gastric bypass surgery. A gastroduodenoscopy with biopsy of the lower duodenum will be performed before the first pharmacokinetic study period.
  Interventions: Drug: paracetamol; Drug: amoxicillin; Drug: talinolol; Procedure: gastroduodenoscopy with biopsy
- post OP (Experimental): The subjects will be administered 200 mg paracetamol, 250 mg amoxicillin and 50 mg talinolol dissolved in 40 ml water which must be drunken with additional 200 ml water on the first study day. This pharmacokinetic period will be performed 5-7 days after the scheduled proximal Roux-en-Y gastric bypass surgery. A sampling of a tissue specimen from the jejunum will be collected during the operation.
  Interventions: Drug: paracetamol; Drug: amoxicillin; Drug: talinolol; Procedure: proximal Roux-en-Y gastric bypass
- one year post OP (Experimental): The subjects will be administered 200 mg paracetamol, 250 mg amoxicillin and 50 mg talinolol dissolved in 40 ml water which must be drunken with additional 200 ml water on the first study day. This pharmacokinetic period and a gastrojejunoscopy with biopsy of the jejunum will be performed about one year after the scheduled proximal stomach bypass surgery.
  Interventions: Drug: paracetamol; Drug: amoxicillin; Drug: talinolol; Procedure: gastrojejunoscopy with biopsy

INTERVENTIONS:
Drug: paracetamol — Administration of 5 ml Paracetamol Saft Hexal (= 200 mg paracetamol)
  Other Names: Paracetamol Saft Hexal
Drug: amoxicillin — Administration of 5 ml Amoxypen® 250 mg Saft (= 250 mg amoxicillin)
  Other Names: Amoxypen® 250 mg Saft
Drug: talinolol — Administration of 1 tablet Cordanum® 50 (= 50 mg talinolol) dissolved with 40 ml tap water
  Other Names: Cordanum® 50
Procedure: gastroduodenoscopy with biopsy — Gastroduodenoscopy with biopsy of the lower duodenum before the first pharmacokinetic study period
  Arms: pre OP
Procedure: gastrojejunoscopy with biopsy — Gastrojejunoscopy with biopsy of the jejunum about one year after proximal Roux-en-Y gastric bypass
  Arms: one year post OP
Procedure: proximal Roux-en-Y gastric bypass — sampling of a tissue specimen from the jejunum during the operation
  Arms: post OP

SUMMARY:
The purpose of this study is to evaluate pharmacokinetics of paracetamol, amoxicillin and talinolol in morbid adipose subjects before as well as shortly after and about one year after proximal Roux-en-Y Gastric Bypass (RYGB) and to measure messenger ribonucleic acid (mRNA) expression and protein content of duodenal and/or jejunal drug metabolizing enzymes (eg. cytochrome P450 isoenzyme 3A4 (CYP3A4), uridine diphosphoglucuronosyltransferase (UGTs)) and drug transport proteins (e.g. P-glycoprotein, MRP2, OATPB, PEPT) before and during the operation and about one year after proximal RYGB.

DETAILED DESCRIPTION:
Intestinal drug absorption appears to be a very complex process characterized by gastrointestinal transit, disintegration of dosage forms, drug dissolution within the intestinal lumen, active and passive uptake processes, mucosal metabolism (e.g. by cytochrome P450 (CYP), UGT, sulfotransferase (SULT) enzymes) and efflux transport by several adenosine triphosphate binding cassette (ABC) transporters as P-glycoprotein, multidrug resistance associated protein (MRP) 2 or breast cancer resistance protein (BCRP). Along the gastrointestinal tract, the upper small intestine (i.e. duodenum, proximal jejunum) represents the main site for absorption of nutrients and drugs offering an appropriately large absorption area of nearly 200 m². Within this bowel segment, there is a high expression of several physiological relevant uptake carriers for nutrients as carbohydrates (e.g. GLUTs), fatty acids (MCTs, FATs), peptides (PEPTs), sterols (NPC1L1) and bile acids (ASBT) which are exclusively located in the small intestine. Furthermore, it is now well established that there is a high intestinal expression of phase I & II metabolizing enzymes as well as drug efflux transporters being responsible for the high first-pass metabolism of many compounds like cyclosporine, nifedipine, midazolam or statins. Apparently, there is a distinct expression gradient along the small intestine (e.g. decreasing levels of P-gp and CYP3A4 but increasing for MRP2). On the other side, the colon features only negligible amounts of enzymes and active uptake and elimination carriers. Therefore, the extent of drug absorption from the bowel is mainly dependent on the intestinal site of drug liberation and, thus, dependent on the administered dosage form, the physicochemical properties of the drug and the individual physiological conditions.

Due to the fact, that under physiological circumstances there is only a low expression of P-gp in the upper parts of the gut (i.e. duodenum and jejunum), a functional "absorption window" is created which enables the preferable absorption of drugs in these proximal region of the small intestine. This is also supported by the markedly higher surface area of the upper small intestine compared to distal segments. It was shown that cyclosporine and talinolol were increasingly less absorbed when delivered into deeper regions of the human intestine. Since both compounds are well established P-gp substrates, this site-dependent absorption phenomenon seems to be caused by the decreasing expression levels of intestinal P-gp counteracting drug uptake into enterocytes. Additionally, it was reported that the effective permeability of atenolol, metoprolol, cimetidine and furosemide was markedly lower in the ileum compared to the jejunum in healthy subjects. These data verified that drug absorption in the lower intestine is less effective than in upper parts which seems to be of outstanding relevance for compounds with predominately duodenal and jejunal absorption (fast release dosage form) and P-gp substrates as ß-lactam antibiotics, furosemide, cyclosporine, talinolol and digoxin.

Consequently, in subjects after massive dissection of the proximal small intestine or after Roux-en-Y gastric bypass surgery, absence of this main intestinal absorption area leads to malabsorption of nutrients (e.g. protein, fat soluble vitamins, minerals and trace elements as iron) and is expected to affect the oral bioavailability of drugs with "absorption window" in the proximal small intestine.

Roux-en-Y gastric bypass surgery, by which the stomach, the duodenum and parts of the jejunum are dislocated from the continuous intestinal passage of the chyme, is the surgical gold standard option to treat morbid adipositas. The method was shown to reduce significantly body weight and obesity-related co-morbidity. Today, this surgical intervention is the most frequently used bariatric surgery (USA: approximately 150.000/year) and its application is still increasing.

Despite its widely use and the well documented risk of nutrient deficiencies, only very little is known about the pharmacokinetic consequences and intestinal adaptation mechanisms in these patients who are often subjected to multiple drug therapy. It was assumed that the reduced intestinal surface area and the reduced time to drug disintegration and dissolution caused by accelerated intestinal transit in these patients are associated with lowered intestinal drug absorption. Additionally, this could be affected by the reduced production of gastric hydrochloric acid by lowering the solubility in case of alkaline drugs. However, it is possible that compensatory processes by other bowel segments could improve drug absorption which could mean that drugs are still adequately absorbed.

From patients with resection of lower intestinal segments (i.e. distal jejunum, ileum, colon) in consequence of Crohn´s disease or ulcerative colitis, the so-called small bowel syndrome, it is known that the pharmacokinetics of drugs as digoxin, cyclosporine, cimetidine and levothyroxine is markedly influenced in form of distinctly reduced intestinal absorption. Furthermore, it was assessed that time-dependent adaptation processes occur in these patients to compensate for the lost of function of the dissected tissue. Therefore, the dependency on parenteral nutrition is decreasing or even full intestinal autonomy will occur. The variety of changes is complex and dependent on the status of the underlying disease, the existing surface area and its functional integrity. These complex adaptation processes are caused by many growth factors, cytokines and hormones (e.g. peptide tyrosine tyrosine (YY), insulin like growth factor (IGF), epidermal growth factor (EGF), glucagon-like peptide (GLP-2), NT).

Most data on adaptive processes in the gastrointestinal tract after dissection of intestinal segments are obtained in animal experiments. These data, however, are not predictive for the situation in man. With regard to the situation after Roux-en-Y gastric bypass surgery, there is no information on how drugs are absorbed after bypassing the stomach, duodenum and parts of the jejunum.

Therefore, pharmacokinetics of three probe drugs (talinolol, paracetamol and amoxicillin) and intestinal expression of intestinal drug metabolizing enzymes (eg. CYP3A4, UGTs) and drug transport proteins (eg. P-gp, MRP2, OATPB, PEPT) before, shortly after (7 days) and one year after the gastric and intestinal bypass surgery in patients with morbid adipositas will be measured. Paracetamol (acetaminophen) was chosen because it is rapidly and completely absorbed from all parts of the gut. Appearance in blood describes the site of drug dissolution within the intestine. Talinolol represents a well established P-gp substrate which absorption is limited by this multidrug transporting protein. Finally, amoxicillin acts as a probe drug for active uptake which is mediated by the peptide transporter PEPT which is predominately expressed in the small intestine and responsible for active H+-coupled uptake of ß-lactam antibiotics and ACE inhibitors.

It is hypothesized that bioavailability of talinolol and amoxicillin will be significantly decreased after the Roux-en-Y gastric bypass surgery compared to the situation before surgery. One year after the surgical intervention, adaptation processes in expression of drug metabolizing enzymes and drug transporters are expected which at least in part compensate for the decrease in bioavailability of the probe drugs.

ELIGIBILITY:
Inclusion Criteria:

* patients who are subjected to proximal stomach-bypass surgery by entire medical reasons independent of the objectives of this study
* age: over 18 years
* sex: male and female
* ethnic origin: Caucasian
* written informed consent

Exclusion Criteria:

* abnormal low hemoglobin values (< 6.5 mmol/l [female]; < 7.6 mmol/l [male])
* obstructive lung disease (e.g. bronchial asthma)
* acute myocardial infarction
* peripheral arterial circulatory disturbance
* any disturbance of impulse formation and conduction
* bradycardia (< 50 beats/min)
* hypotension (systolic pressure < 90 mmHg)
* phaeochromocytoma
* subjects who are unable to understand the written and verbal instructions, in particular regarding the risks and inconveniences they will be exposed to as a result of their participation in the study
* blood donation or other blood loss of more than 400 ml within the last 3 months prior to the start of the study
* participation in a clinical trial during the last 3 months prior to the start of the study
* less than 14 days after last acute disease
* treatment with paracetamol, amoxicillin or talinolol 7 days before the study
* repeated use of drugs during the last 4 weeks prior to the intended first administration, which can influence drug biotransformation and drug transport
* intake of grapefruit containing food or beverages within 7 days prior to administration
* known allergic reactions to the active ingredients used or to constituents of the pharmaceutical preparation, also against penicillin
* subjects with severe allergies or multiple drug allergies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-06; Primary Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
area under the concentration time curve of paracetamol, amoxicillin and talinolol | up to 1.5 h before and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24 h after study medication

SECONDARY OUTCOMES:
maximal concentration of the concentration time curve of paracetamol, amoxicillin and talinolol | up to 1.5 h before and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24 h after study medication
timepoint of the maximal concentration of the concentration time curve of paracetamol, amoxicillin and talinolol | up to 1.5 h before and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24 h after study medication
terminal half-life of the concentration time curve of paracetamol, amoxicillin and talinolol | up to 1.5 h before and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24 h after study medication
mRNA expression determined by quantitative polymerase chain reaction given as cycle threshold normalized to house keeping gene 18S and villin | up to 2 days before the first study medication and after at least 6 h fasting, during proximal Roux-en-Y gastric bypass surgery within 3 days after first study medication and about one year after proximal Roux-en-Y gastric bypass surgery
  mRNA expression of duodenal and/or jejunal drug metabolizing enzymes (eg. CYP3A4, UGTs) and drug transport proteins (e.g. P-glycoprotein, MRP2, OATPB, PEPT)
protein abundance determined by liquid chromatography-mass spectrometry based targeting proteomics normalized to villin | up to 2 days before the first study medication and after at least 6 h fasting, during proximal Roux-en-Y gastric bypass surgery within 3 days after first study medication and about one year after proximal Roux-en-Y gastric bypass surgery
  protein content of duodenal and/or jejunal drug metabolizing enzymes (eg. CYP3A4, UGTs) and drug transport proteins (e.g. P-glycoprotein, MRP2, OATPB, PEPT)

CONTACTS AND LOCATIONS:
Overall Officials: Werner Siegmund, Prof, Principal Investigator — Department of Clinical Pharmacology
Locations (2):
- Germany (2):
  - Department of Clinical Pharmacology, Ernst-Moritz-Arndt-University Greifswald, Greifswald, Mecklenburg-Vorpommern
  - Surgical Clinic of the Clinical Centre Suedstadt Rostock, Rostock